CLINICAL TRIAL: NCT02808650
Title: A Phase 1 Study of LY2606368 (Prexasertib Mesylate Monohydrate) a CHK1/2 Inhibitor, in Pediatric Patients With Recurrent or Refractory Solid Tumors, Including CNS Tumors
Brief Title: Prexasertib in Treating Pediatric Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1515; NCI-2016-00643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1515; ADVL1515 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1515 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Childhood Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Primary Central Nervous System Neoplasm; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (prexasertib) (Experimental): Patients receive prexasertib IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacokinetic (PK) study; Drug: Prexasertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacokinetic (PK) study — Correlative studies
Drug: Prexasertib — Given IV
  Other Names: LY2606368

SUMMARY:
This phase I trial studies the side effects and best dose of prexasertib in treating pediatric patients with solid tumors that have come back after a period of time during which the tumor could not be detected or does not respond to treatment. Checkpoint kinase 1 inhibitor LY2606368 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of prexasertib (LY2606368) administered as an intravenous (IV) infusion over 60 minutes, every 14 days of a 28-day cycle to children with recurrent or refractory solid tumors.

II. To define and describe the toxicities of LY2606368 administered on this schedule.

III. To characterize the pharmacokinetics of LY2606368 in children with recurrent or refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of LY2606368 within the confines of a phase 1 study.

II. To examine checkpoint kinase (CHK)1/2 expression status in archival tumor tissue from solid tumor pediatric patients using immunohistochemistry.

III. To evaluate tumor tissue for deletion and/or mutation of tumor protein 53 (TP53) as a potential biomarker of Chk1 inhibition.

IV. To evaluate autophosphorylation of Chk1 and H2A histone family, member x (H2AX) in peripheral blood mononuclear cells as a potential pharmacodynamic marker of LY2606368 activity.

OUTLINE: This is a dose-escalation study.

Patients receive prexasertib IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or refractory solid tumors, including central nervous system (CNS) tumors, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or in patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 % for patients =< 16 years of age

  * Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the defined eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days must have elapsed from last dose of agent; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days must have elapsed since the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days must have elapsed since the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days must have elapsed after infusion, and no evidence of graft-versus-host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days must have elapsed after completion
  * Cellular therapy: >= 42 days must have elapsed since the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * X ray (XRT)/external beam irradiation including protons: >= 14 days must have elapsed after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131 iodine metaiodobenzylguanidine [131I-MIBG]): >= 42 days must have elapsed since systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to LY2606368
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin >= 8.0 g/dl at baseline (may receive packed red blood cell [PRBC] transfusions)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: maximum serum creatinine (mg/dL)
  * 1 to < 2 years: 0.6 (male and female)
  * 2 to < 6 years: 0.8 (male and female)
  * 6 to < 10 years: 1 (male and female)
  * 10 to < 13 years: 1.2 (male and female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (3x ULN); for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
* Corrected QT (QTc) =< 480 msec

  * Note: Patients should avoid concomitant medication known or suspected to prolong QTc interval or cause Torsades De Pointes; If possible, alternative agents should be considered
  * Patients who are receiving drugs that prolong the QTc are eligible if the drug is necessary and no alternatives are available
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v]4) resulting from prior therapy must be =< grade 2
* For patients with CNS tumors, any baseline neurologic deficit, including seizures, must be stable for at least one week prior to initiating study treatment
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent if available; if tissue blocks or slides are unavailable, the study chair must be notified prior to study enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method both during and for 3 months after participation in this study; abstinence is an acceptable method of contraception
* Corticosteroids: Patients receiving corticosteroids must have been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible
* Anti-GVHD agents post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Strong CYP1A2 inhibitors: Patients must not have received strong CYP1A2 inhibitors (ciprofloxacin, fluvoxamine, zafirlukast) for at least 7 days prior to enrollment and must not receive them for the duration of the study
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to LY2606368 or to its formulation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Wetmore, Principal Investigator — COG Phase I Consortium
Locations (21):
- United States (21):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Cash T, Fox E, Liu X, Minard CG, Reid JM, Scheck AC, Weigel BJ, Wetmore C. A phase 1 study of prexasertib (LY2606368), a CHK1/2 inhibitor, in pediatric patients with recurrent or refractory solid tumors, including CNS tumors: A report from the Children's Oncology Group Pediatric Early Phase Clinical Trials Network (ADVL1515). Pediatr Blood Cancer. 2021 Sep;68(9):e29065. doi: 10.1002/pbc.29065. Epub 2021 Apr 21. PMID 33881209

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Dose Level 1: 80 mg/m^2; Part A Dose Level 2: 100 mg/m^2; Part A Dose Level 3: 125 mg/m^2; Part A Dose Level 4: 150 mg/m^2; Part PK Dose Level 4: 150 mg/m^2: Patients receive prexasertib IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Started | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 5 | 5 | 6 | 5 | 4
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 4 | 4 | 6 | 25
  Between 18 and 65 years | 0 | 1 | 2 | 2 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8.5 [2.0 to 17.0] | 14 [4.0 to 20.0] | 10 [3.0 to 19.0] | 16.5 [7.0 to 20.0] | 4.5 [3.0 to 13.0] | 9.5 [2.0 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 6 | 9
  Male | 6 | 4 | 5 | 6 | 0 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 2 | 5
  Not Hispanic or Latino | 6 | 3 | 5 | 6 | 4 | 24
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 1 | 3
  White | 5 | 4 | 2 | 6 | 3 | 20
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 3 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Prexasertib
Description: Maximum tolerated dose or recommended phase 2 dose of prexasertib assessed by national Cancer Institute (NCI) CTCAE version 4.0 defined as the maximum dose at which fewer that one-third of patients experience a dose limiting toxicity in cycle 1
Time Frame: Up to 28 days
Measure: Number; unit: mg/m^2
Arm/Group | Treatment (Prexasertib)
Number analyzed (Participants) | 25
mg/m^2 | 150

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) to Prexasertib
Description: Number of patients with DLT to Prexasertib by dose level and study part.
Time Frame: Up to 28 days
Population: All Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Area Under the Concentration Time Curve for Prexasertib
Description: Median (min, max) area under the concentration by time curve for prexasertib assessed at 1, 1.5, 2, 4, and 8 hours on day 1 post infusion by dose level and study part
Time Frame: Up to 8 hours
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*ng/mL | 1718.7 [1215.2 to 2168.6] | 2285.5 [1658.4 to 3529.0] | 2534.4 [2080.0 to 3535.6] | 4206.6 [2164.9 to 5357.9] | 3097.7 [2443.2 to 4282.5]

4. Secondary Outcome: Antitumor Activity of Prexasertib
Description: Number of response evaluable patients with response (CR/PR) using the RECIST guideline version 1.1 including CR: disappearance of all target and non-target lesions; PR: at least 30% decrease in the sum of the diameters of target lesions by dose level and study part
Time Frame: Up to 2 years
Population: Eligible Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: CHK1/2 Expression Status
Description: Number of patients with CHK1/2 expression by percent of tumor cells with CHK1/2 expression defined by quartiles.
Time Frame: Up to 2 years
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 6 | 1 | 3 | 5 | 4
Participants
  0% Negative | 2 | 0 | 1 | 0 | 1
  1-25% cells positive | 0 | 0 | 0 | 1 | 1
  26-50% cells positive | 1 | 0 | 1 | 0 | 0
  51-75% cells positive | 2 | 0 | 1 | 1 | 2
  76-100% cells positive | 1 | 1 | 0 | 3 | 0

6. Secondary Outcome: TP53 Deletion and/or Mutation in Tumor Tissue as a Potential Biomarker of Chk1 Inhibition
Description: Number of patients with TP53 deletion and/or mutation of Trp53 by percent of tumor cells with TP53 deletion and/or mutation of Trp53 defined by quartiles.
Time Frame: Up to 2 years
Population: Response evaluable Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 6 | 1 | 3 | 5 | 4
Participants
  0% Negative | 1 | 0 | 1 | 0 | 0
  1-25% cells positive | 0 | 0 | 0 | 2 | 1
  26-50% cells positive | 1 | 1 | 0 | 0 | 0
  51-75% cells positive | 2 | 0 | 1 | 1 | 0
  76-100% cells positive | 2 | 0 | 1 | 2 | 3

7. Secondary Outcome: Autophosphorylation of CHK1 and H2AX
Description: Median (min, max) autophosphorylation of CHK1 and H2AX in peripheral blood mononuclear cells by dose level and study part.
Time Frame: Up to 2 years
Population: Testing failed. Data not available to be reported for outcome measure.
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Part A Dose Level 1: 80 mg/m^2 | Part A Dose Level 2: 100 mg/m^2 | Part A Dose Level 3: 125 mg/m^2 | Part A Dose Level 4: 150 mg/m^2 | Part PK Dose Level 4: 150 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/6 | 0/6 | 0/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/6 | 2/6 | 4/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 80 mg/m^2 (N=6) | Part A Dose Level 2: 100 mg/m^2 (N=6) | Part A Dose Level 3: 125 mg/m^2 (N=6) | Part A Dose Level 4: 150 mg/m^2 (N=6) | Part PK Dose Level 4: 150 mg/m^2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 80 mg/m^2 (N=6) | Part A Dose Level 2: 100 mg/m^2 (N=6) | Part A Dose Level 3: 125 mg/m^2 (N=6) | Part A Dose Level 4: 150 mg/m^2 (N=6) | Part PK Dose Level 4: 150 mg/m^2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Abducens nerve disorder (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0 | 1 | 2
Agitation (Psychiatric disorders) | 2 | 2 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 3 | 2 | 0 | 3
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 6 | 4 | 6 | 5
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 3 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 1 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 2 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 3 | 1
Blood and lymphatic system disorders - Other, DECREASED RED BLOOD CELL (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0
Cardiac disorders - Other, DIFFUSE T WAVE CHANGE (POST TREATEMENT EKG) (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, DIFFUSED T WAVE CHANGES (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, EJECTION MURMUR (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 3 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3 | 3
Creatinine increased (Investigations) | 0 | 0 | 2 | 2 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 4 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 | 2 | 3 | 2 | 3
Endocrine disorders - Other, DEVELOPMENTAL DELAY (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Endocrine disorders - Other, GROWTH FAILURE; HX OF PRECOCIOUS PUBERTY; ADVANCED BONE AGE (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, AMBLYOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, EXOTROPIA (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, LAGOPHTHALMOS (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, R PUPIL LARGER THAN L AND LESS REACTIVE (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 2 | 1 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 4 | 4 | 5 | 4
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Fever (General disorders) | 3 | 1 | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 2 | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, NODULAR LOCALIZED EDEMA (General disorders) | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, NODULAR/LOCALIZED EDEMA (General disorders) | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Growth hormone abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 3 | 4
Hearing impaired (Ear and labyrinth disorders) | 2 | 1 | 1 | 1 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1
Hepatobiliary disorders - Other, BILIARY DRAIN (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 3 | 3 | 2 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 3
Hypoglossal nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 1 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 3 | 3 | 1 | 4
Hypotension (Vascular disorders) | 2 | 0 | 1 | 1 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0 | 0
IVth nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Immune system disorders - Other, SEASONAL ALLERGIES (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, COLON (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (General disorders) | 1 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 1 | 4 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Investigations - Other, ALKALINE PHOSPHATASE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, ANION GAP INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE LOW (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, DECREASED ALK PHOS (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, DECREASED BLOOD OSMOLALITY (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, DECREASED CO2 (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 0 | 0 | 1 | 0
Investigations - Other, ELEVATED CRP (Investigations) | 1 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, HYPERAMMONEMIA (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, HYPERCHLOREMIA (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, INCREASED CRP (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, SERUM BICARBONATE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 3 | 4 | 4 | 3
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition disorders - Other, DECREASED CHLORIDE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, INCREASED CHLORIDE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SCIATIC PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, INTRATUMORAL HEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, LEFT LOWER POSTERIOR FO (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, ABNORMAL BALANCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, DYSMETRIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, INTRA-TUMORAL HEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, SEIZURE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, TWITCHING (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 6 | 6 | 5 | 6 | 6
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 2 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 3 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 2 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 4 | 6 | 5 | 4 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Psychiatric disorders - Other, ADHD (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, HYPERINFLATED CHEST (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, SHALLOW BREATHING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 2 | 4 | 3 | 3
Skin and subcutaneous tissue disorders - Other, COLD SORE PRESUMED HSV INFECTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, EYELID RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, INGROWING TOENAIL (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PLANTAR WART (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ULCER/SKIN BREAKDOWN TO RIGHT ELBOW (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 2 | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Surgical and medical procedures - Other, BILIARY CATHETER REPLACEMENT (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Surgical and medical procedures - Other, ELECTIVE TUMOR RESECTION (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, SHUNT MALFUNCTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 1 | 3 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Vagus nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 2 | 3 | 4
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0
Weight loss (Investigations) | 2 | 2 | 1 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 6 | 6 | 5 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT02808650/Prot_SAP_000.pdf